CLINICAL TRIAL: NCT04119661
Title: Postendodontic Pain on Using Max-i-Probe vs NaviTip as Irrigation Needles: A Randomized Clinical Trial
Brief Title: Postendodontic Pain on Using Max-i-Probe vs NaviTip as Irrigation Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzan AW Amin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENDO-CU-2012-7-15
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Max-i-Probe (Experimental)
  Interventions: Device: Max-i-Probe
- NaviTip (Active Comparator)
  Interventions: Device: NaviTip

INTERVENTIONS:
Device: Max-i-Probe — Using Max-i-Probe as endodontic needle during syringe irrigation
  Arms: Max-i-Probe
Device: NaviTip — Using NaviTip as endodontic needle during syringe irrigation
  Arms: NaviTip

SUMMARY:
The aim of this prospective, randomized, clinical trial was to evaluate the effect of the side-vented Max-i-Probe versus the end-vented NaviTip as endodontic needles during syringe irrigation on post-operative pain in adult patients with symptomatic irreversible pulpitis in posterior mandibular teeth.

DETAILED DESCRIPTION:
The aim of this prospective, randomized, clinical trial was to evaluate the effect of the side-vented Max-i-Probe versus the end-vented NaviTip as endodontic needles during syringe irrigation on post-operative pain in adult patients with symptomatic irreversible pulpitis in posterior mandibular teeth. Medical and dental history was obtained from all participants in this trial and clinical examination for teeth was performed. Participants with symptomatic irreversible pulpitis were included. After access cavity preparation, participants were randomly assigned to one of the following groups: experimental group (Max-i-Probe) or control group (NaviTip). One-visit root canal treatment was performed . Each patient received a 48-h diary to record postoperative pain. Post-operative pain was measured at the following time points: 4, 12, 24 and 48 hours after root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 16-65 year old.
2. Medically free.
3. Mandibular posterior teeth with symptomatic irreversible pulpitis.
4. No sex predilection

Exclusion Criteria:

1. Pregnant females.
2. History of allergy to any medication used in the study.
3. Preoperative premedication less than 6 hours before procedure.
4. Cracked teeth and teeth with badly-decayed crowns.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain using a pain-measuring scale | 4 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 4h after root canal treatment
Postoperative pain using a pain-measuring scale | 12 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 12h after root canal treatment
Postoperative pain using a pain-measuring scale | 24 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 24 h after root canal treatment
Postoperative pain using a pain-measuring scale | 48 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 48h after root canal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Amin, Professor, Study Director — Cairo University; Mohamed El-Bayoumi, Professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gondim E Jr, Setzer FC, Dos Carmo CB, Kim S. Postoperative pain after the application of two different irrigation devices in a prospective randomized clinical trial. J Endod. 2010 Aug;36(8):1295-301. doi: 10.1016/j.joen.2010.04.012. Epub 2010 Jun 19. PMID 20647083
- [Background] Middha M, Sangwan P, Tewari S, Duhan J. Effect of continuous ultrasonic irrigation on postoperative pain in mandibular molars with nonvital pulps: a randomized clinical trial. Int Endod J. 2017 Jun;50(6):522-530. doi: 10.1111/iej.12666. Epub 2016 Jun 28. PMID 27248848